CLINICAL TRIAL: NCT07319000
Title: Efficacy of Low-dose Post-transplant Cyclophosphamide for Prevention of Graft-versus-host Disease in Ambulatory Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of Low-dose PT-Cy for Prevention of GVHD in Ambulatory Allogeneic HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Cesar Homero Gutierrez-Aguirre, Professor of Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE22-0037
Record Dates: First submitted 2025-09-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease
Keywords: Transplants; Cyclophosphamide
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: A consecutive sample of 35 patients undergoing allogeneic transplantation will be included and will be administered low-dose post-transplant cyclophosphamide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose post-transplant cyclophosphamide (Experimental): Low dose post-transplant cyclophosphamide therapy will be administered as follows:
  Allogeneic stem cell transplant:
  Cyclophosphamide 30/mg/kg/day for 2 continuous days.
  Haploidentical stem cell transplant:
  Cyclophosphamide 40/mg/kg/day for 2 continuous days.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — low-dose post-transplant cyclophosphamide

SUMMARY:
Low-dose post-transplant cyclophosphamide have demonstrated therapeutic efficacy in allogeneic stem cell transplants which is comparable with the standard dose and also facilitates early hematological recovery.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) is the most important complication that occurs in hematopoietic stem cell transplantation (HSCT). GVHD prophylaxis based on the use of post-transplant cyclophosphamide (PT-Cy) has proven to be a practical, easily and accessible agent that allows both identical and haploidentical transplants to be performed with lower incidences of this disease.

Low-dose cyclophosphamide have already demonstrated therapeutic efficacy in these types of transplants which is comparable with the standard dose and also facilitates early hematological recovery that can in turn reduce risks of infection, hospital stay and total costs for the patient.

The investigators will conduct a phase 2, non-randomized, single center, non-comparative clinical trial to demonstrate the effectiveness of of low-dose PT-Cy which is accessible to a population with limited resources while maintaining acceptable efficacy and safety to prevent GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Both genders.
* Diagnosis of any blood disease in need of an allogeneic bone marrow transplant (aplastic anemia, acute myeloid leukemia, chronic granulocytic leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, chronic myelomonocytic leukemia, Hodgkin lymphoma, and Non-Hodgkin lymphoma).
* Patients who have compatible related donors to perform an identical or haploidentical allogeneic transplant.
* Patients with functional status 0 to 2 using the ECOG scale.

Exclusion Criteria:

* Poor functional status (ECOG>2).
* Organic dysfunction (Marshall score ≥2).
* Pregnancy
* Heart failure (NYHA III or IV).
* Renal failure (GFR <30 ml/min/1.72m2).
* History of ventricular arrhythmias or uncontrolled arrhythmias.
* Acute myocardial infarction, unstable angina, or stable angina in the last six months.
* Uncontrolled active infection.
* Liver disease (Child-Pugh C).
* Patients not approved by the local transplant committee for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of Low-dose PT-Cy | 6 months
  Low-dose PT-Cy (30 and 40 mg/kg/day/2 days) is effective in achieving an incidence of grade III/IV (Glucksberg grade) acute GVHD and moderate to severe chronic GVHD equal to or below historical controls of 20 and 30%, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Monterrey, Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sugita J, Kamimura T, Ishikawa T, Ota S, Eto T, Kuroha T, Miyazaki Y, Kumagai H, Matsuo K, Akashi K, Taniguchi S, Harada M, Teshima T. Reduced dose of posttransplant cyclophosphamide in HLA-haploidentical peripheral blood stem cell transplantation. Bone Marrow Transplant. 2021 Mar;56(3):596-604. doi: 10.1038/s41409-020-01065-0. Epub 2020 Sep 24. PMID 32973350